CLINICAL TRIAL: NCT06054568
Title: Ventricular-arterial Coupling of the Heart Among Patients With Mitral Stenosis Undergoing Percutaneous Trans-luminal Mitral Commissurotomy. Cardiac Magnetic Resonance Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Zakher Bakhiet, assistant lecturer, Assiut University
Other Study IDs: Cardiac magnetic resonance
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-09

CONDITIONS: Mitral Valve Stenosis
Keywords: Mitral stenosis; cardiac magnetic resonance
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Mitral stenosis undergoing Percutaneous Mitral trans-luminal commissurotomy

SUMMARY:
Although the incidence of rheumatic fever and its complications has declined in developed countries, the disease remains a major health problem in many developing countries. It is estimated that up to 30 million school-age children and young adults worldwide suffer from chronic rheumatic heart disease, and almost a third of them suffer from mitral valve stenosis (MS).

Various treatments are currently available to patients, including medical, surgical, and percutaneous mitral commissurotomy (PTMC), depending on the severity of symptoms, the type and severity of mitral stenosis, and the morphology of the mitral valve.

Successfully performed PTMC increases the optimal mitral valve area and is unlikely to result in significant mitral valve regurgitation. PTMC candidates are selected according to the latest European society of cardiology (ESC) guidelines for the treatment of mitral stenosis based on echocardiographic examination of the mitral valve and its dimensions. The Wilkins score, determined using ultrasound, is an important tool for patient selection.

CMR provides tomographic assessment of the heart with high spatial resolution and enables accurate assessment of ventricular volume, identification of segmental kinetic abnormalities, and detection of tissue changes such as fibrosis, edema, or fatty substitution.

Patients with severe mitral stenosis who underwent percutaneous mitral commissurotomy (PTMC) showed significant changes in right ventricular (RV) function. One study assessed the pre and post changes in RV function after PTMC and found significant improvements in RV parameters such as RV systolic pressure, RV outlet FS, RV TEi index, RV wall thickness, and pulmonary artery systolic pressure.

Successful balloon mitral valvuloplasty (BMV) in patients with rheumatic mitral stenosis (MS) is associated with improvement in left ventricular (LV) function and remodeling. A study using cardiac magnetic resonance imaging (CMR) found that BMV led to an increase in LV peak systolic global longitudinal strain (GLS) and global circumferential strain (GCS) at 6 months, with further improvement at 1 year.

Ventriculo-arterial coupling (VAC) plays an important role in the physiology of cardiac and aortic mechanics as well as in the pathophysiology of heart disease. VAC assessment has independent diagnostic and prognostic value and can be used to improve risk stratification and monitor therapeutic interventions. Traditionally, VAC is assessed by noninvasive measurement of the end-systolic elasticity ratio of arteries (Ea) and ventricles (Ees). Therefore, measuring any component of this ratio or new, more sensitive myocardial markers (e.g.B. global longitudinal strain) and arterial function (e.g. pulse wave velocity) can better characterize the VAC. In valvular heart disease, systemic arterial compliance and valve-arterial impedance have established diagnostic and prognostic value and can monitor the effects of valve replacement on vascular and cardiac function. Treatment to improve VAC by improving one of its components may delay the onset of heart failure and potentially improve the prognosis of heart failure.

According to Ozdogru I et al, A study of patients with severe mitral stenosis undergoing percutaneous balloon valvuloplasty and healthy subjects, demonstrated that mitral stenosis induced an increase in arterial stiffness that was improved after percutaneous balloon valvuloplasty.

Diastolic dysfunction has emerged as an important predictor of adverse outcomes in multiple forms of congenital heart disease.

A recently derived CMR prognostic tool, the left atrioventricular coupling index (LACI), has been evaluated as part of the Multi-Ethnic Study of Atherosclerosis (MESA). LACI is defined as the ratio between LA end-diastolic volume and LV end diastolic volume. It was created to determine whether the close physiological relationship between the LA and LV could serve as a primary prevention tool in the early detection of cardiovascular disease. LACI has been shown to serve as a strong predictor for the incidence of heart failure, atrial fibrillation, cardiovascular disease, and coronary heart disease death in healthy adult populations. A novel right atrioventricular coupling index can potentially help with risk stratification, novel parameter, termed the Right Atrioventricular Coupling Index (RACI), and was defined as the ratio of RA end-diastolic volume to right ventricle (RV) end-diastolic volume.

According to our knowledge there was no specific study was done using cardiac magnetic resonance imaging (CMR) for assessment of Ventricular-arterial coupling pre and post PTMC

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe MS eligible for PTMC according to the recent ESC Guidelines for the management of valvular heart disease 2021

Exclusion Criteria:

1. Patient with contraindication to CMR (e.g. due to pacemakers, implantable cardioverter defibrillators, claustrophobia, .. etc)
2. Patients with associated coronary artery disease.
3. Patients with other significant valvular heart disease including organic tricuspid valve disease
4. Patients with any type of cardiomyopathy
5. Patients with renal impairment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with mitral stenosis undergoing PTMC
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of atrio-ventricular coupling and ventricular arterial coupling assessed via cardiac magnetic resonance pre and post percutaneous trans-luminal mitral commissurotomy at the pre-specified time points | 1 year

IPD SHARING:
Plan to Share IPD: Undecided
because it not decided till now

REFERENCES:
- [Background] Ikonomidis I, Aboyans V, Blacher J, Brodmann M, Brutsaert DL, Chirinos JA, De Carlo M, Delgado V, Lancellotti P, Lekakis J, Mohty D, Nihoyannopoulos P, Parissis J, Rizzoni D, Ruschitzka F, Seferovic P, Stabile E, Tousoulis D, Vinereanu D, Vlachopoulos C, Vlastos D, Xaplanteris P, Zimlichman R, Metra M. The role of ventricular-arterial coupling in cardiac disease and heart failure: assessment, clinical implications and therapeutic interventions. A consensus document of the European Society of Cardiology Working Group on Aorta & Peripheral Vascular Diseases, European Association of Cardiovascular Imaging, and Heart Failure Association. Eur J Heart Fail. 2019 Apr;21(4):402-424. doi: 10.1002/ejhf.1436. Epub 2019 Mar 12. PMID 30859669
- [Background] Samaan AA, Said K, Aroussy WE, Hassan M, Romeih S, El Sawy A, Fawzy ME, Yacoub M. Left Ventricular Remodeling Following Balloon Mitral Valvuloplasty in Rheumatic Mitral Stenosis: Magnetic Resonance Imaging Study. Front Cardiovasc Med. 2021 Jun 4;8:674435. doi: 10.3389/fcvm.2021.674435. eCollection 2021. PMID 34150869
- [Background] Muhammad, Abdul, Wahab., Syed, Aziz-Ur, Rahman., Umer, Shafiq. (2022). Effect of percutaneous transvenous mitral commisurotomy (ptmc) on right ventricular function. Pakistan Heart Journal, 55(Supplement1):S13-S13. doi: 10.47144/phj.v55isupplement1.2429
- [Background] Alec Vahanian, Friedhelm Beyersdorf, Fabien Praz, Milan Milojevic, Stephan Baldus, Johann Bauersachs, Davide Capodanno, Lenard Conradi, Michele De Bonis, Ruggero De Paulis, Victoria Delgado, Nick Freemantle, Martine Gilard, Kristina H Haugaa, Anders Jeppsson, Peter Jüni, Luc Pierard, Bernard D Prendergast, J Rafael Sádaba, Christophe Tribouilloy, Wojtek Wojakowski, ESC/EACTS Scientific Document Group , ESC National Cardiac Societies , 2021 ESC/EACTS Guidelines for the management of valvular heart disease: Developed by the Task Force for the management of valvular heart disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS), European Heart Journal, Volume 43, Issue 7, 14 February 2022, Pages 561-632, https://doi.org/10.1093/eurheartj/ehab395
- [Background] Stefanadis C, Stratos C, Pitsavos C, Kallikazaros I, Triposkiadis F, Trikas A, Vlachopoulos C, Gavaliatsis I, Toutouzas P. Retrograde nontransseptal balloon mitral valvuloplasty. Immediate results and long-term follow-up. Circulation. 1992 May;85(5):1760-7. doi: 10.1161/01.cir.85.5.1760. PMID 1572032
- [Background] Seckeler MD, Hoke TR. The worldwide epidemiology of acute rheumatic fever and rheumatic heart disease. Clin Epidemiol. 2011 Feb 22;3:67-84. doi: 10.2147/CLEP.S12977. PMID 21386976